CLINICAL TRIAL: NCT03765671
Title: An Open-label, Phase 1, Single-dose Study to Evaluate the Pharmacokinetics of Elafibranor 120 mg in Adult Subjects With Hepatic Impairment and Adult Healthy Control Subjects
Brief Title: Elafibranor Pharmacokinetic Parameters in Hepatic Impaired Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genfit (Industry)
Collaborators: Syneos Health (Other); University of Miami (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GFT505-118-14
Record Dates: First submitted 2018-11-30; First posted 2018-12-05 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Hepatic Impairment; Liver Disease; Pharmacokinetics
MeSH Terms: conditions — Liver Diseases | interventions — 2-(2,6-dimethyl-4-(3-(4-(methylthio)phenyl)-3-oxo-1-propenyl)phenoxyl)-2-methylpropanoic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Mild Child-Pugh A (Experimental): Single oral dose of elafibranor 120mg
  Interventions: Drug: Elafibranor
- Moderate Child-Pugh B (Experimental): Single oral dose of elafibranor 120mg
  Interventions: Drug: Elafibranor
- Severe Child-Pugh C (Experimental): Single oral dose of elafibranor 120mg
  Interventions: Drug: Elafibranor
- Healthy (Experimental): Single oral dose of elafibranor 120mg
  Interventions: Drug: Elafibranor

INTERVENTIONS:
Drug: Elafibranor — 120mg oral single dose
  Other Names: GFT505

SUMMARY:
This study is being conducted in order to assess the need for dose adjustment for elafibranor in patients with hepatic impairment. Pharmacokinetic parameters of elafibranor and its active metabolite (GFT1007) will be compared in hepatic impaired patients (mild, moderate and severe according to Child-Pugh categories) versus healthy participants after a single oral administration of elafibranor 120 mg.

ELIGIBILITY:
Inclusion Criteria:

- For all participants:

1. Males or females, between 18 and 75 years of age, inclusive;
2. With a minimum body weight of 50 kg and within a BMI range of 18.0 to 40.0 kg/m², inclusive;
3. Females participating in this study must be of non-childbearing potential or using highly efficient contraception for the full duration of the study
4. Negative serum pregnancy test at screening (if applicable);
5. Negative human immunodeficiency virus antibody screens at Screening;

   * For hepatically impaired participants:
6. Participants who have chronic (≥ 6 months) mild, moderate, or severe hepatic insufficiency (of any etiology) that has been clinically stable (no acute episodes of illness due to deterioration in hepatic function) for at least 1 month prior to Screening Currently on a stable medication regimen

   * For healthy volunteers with normal hepatic function:
7. Non-smokers
8. Matched to participants with Mild and/or Moderate and/or Severe hepatic impairment in age (± 10 years), BMI (± 20 percent) and gender.

Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

- For all participants:

1. A positive alcohol test result at Check-in;
2. A history of alcohol abuse in the prior 2 years;
3. Positive urine screen for drugs of abuse at Screening or Check-in.
4. Strenuous exercise within 72 hours prior to Check-in;
5. Blood donation or loss of blood (excluding volume drawn at screening or menses) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to the dosing;
6. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs except that appendectomy and hernia repair will be allowed. Bariatric surgery will not be allowed.
7. Presence or history of malignancy within the prior 3 years, with the exception of treated basal cell or squamous cell carcinoma;
8. Poor peripheral venous access;
9. Receipt of blood products within 2 months prior to Check-in;

   * For hepatically impaired participants:
10. History of unstable diabetes mellitus Subjects who have a transjugular intrahepatic portosystemic shunt and/or have undergone portacaval shunting;
11. Participant has shown evidence of hepatorenal syndrome or has creatinine clearance ≤ 60 mL/min Subject has required treatment for GI bleeding within the 6 months prior to Check in;
12. Recent history of paracentesis (< 3 months prior to Check-in);
13. Participants with Wilson's disease, alpha-1 antitrypsin deficiency, glycogen storage diseases, or galactosemia;
14. Participants with anemia secondary to hepatic disease, unless hemoglobin is ≥ 9 g/dL and anemia symptoms are not clinically significant. Subjects must have ≥ 35 000 platelets at screening and at Day -1;

    * For healthy volunteers with normal hepatic function:
15. Significant history or clinical manifestation of any metabolic (including thyroid), allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular (including any prior history of cardiomyopathy or cardiac failure), gastrointestinal (GI), neurological, or psychiatric disorder;
16. Positive serologic test for hepatitis B surface antigen or for hepatitis C virus antibody at Screening;
17. Frequent headaches (> twice a month) and/or migraines, recurrent nausea and/or vomiting;
18. Participants with symptomatic hypotension at Screening, whatever the decrease of blood pressure, or asymptomatic postural hypotension;
19. Cholecystectomy

Other protocol-defined exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-06-14 (Actual)

PRIMARY OUTCOMES:
Area under curve from dosing time to last measurement (AUC(0-t)) of elafibranor and active metabolite | pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose. Additionally, after elafibranor administration at 288 and 384 hours for hepatic impaired patients
  In participants with mild, moderate and severe hepatic impairment compared to healthy volunteers
Area under curve from dosing time to infinity (AUC(0-∞)) of elafibranor and active metabolite | pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose. Additionally, after elafibranor administration at 288 and 384 hours for hepatic impaired patients
  In participants with mild, moderate and severe hepatic impairment compared to healthy volunteers

SECONDARY OUTCOMES:
Plasma pharmacokinetics: maximum plasma drug concentration (Cmax) | pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose. Additionally, after elafibranor administration at 288 and 384 hours for hepatic impaired participants
  for elafibranor and metabolites
Plasma pharmacokinetics: elimination half-life (t1/2) | pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose. Additionally, after elafibranor administration at 288 and 384 hours for hepatic impaired participants
  for elafibranor and metabolites
Plasma pharmacokinetics: apparent volume of distribution (Vd/F) | pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose. Additionally, after elafibranor administration at 288 and 384 hours for hepatic impaired participants
  for elafibranor
Plasma pharmacokinetics: renal clearance (CLr) | pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose. Additionally, after elafibranor administration at 288 and 384 hours for hepatic impaired participants
  for elafibranor and metabolites
Plasma pharmacokinetics: apparent non renal clearance (CLnr/F) | pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose. Additionally, after elafibranor administration at 288 and 384 hours for hepatic impaired participants
  for elafibranor
Plasma pharmacokinetics: apparent total clearance (CL/F) | pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose. Additionally, after elafibranor administration at 288 and 384 hours for hepatic impaired participants
  for elafibranor
Plasma pharmacokinetics: area under the plasma concentration-time curve extrapolated from time t to infinity as a percentage of total area under the plasma concentration-time curve (%AUCextra) | pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose. Additionally, after elafibranor administration at 288 and 384 hours for hepatic impaired participants
  for elafibranor and metabolites
Plasma pharmacokinetics: area under curve from dosing time to last measurement (AUC(0-t)) of glucuronide metabolites and corresponding aglycones | pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose. Additionally, after elafibranor administration at 288 and 384 hours for hepatic impaired participants
  for the glucuronide metabolites of elafibranor and corresponding aglycones
Plasma pharmacokinetics: area under curve from dosing time to infinity (AUC(0-∞)) of glucuronide metabolites and corresponding aglycones | pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose. Additionally, after elafibranor administration at 288 and 384 hours for hepatic impaired patients
  for the glucuronide metabolites of elafibranor and corresponding aglycones
Urine pharmacokinetics: amount excreted (Ae) | pre-dose and then 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  for elafibranor and metabolites, if applicable. 24 hours urine collection from dosing to 216 hours post-dose
Urine pharmacokinetics: cumulative amount excreted (Ae0-t) | pre-dose and then 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  for elafibranor and metabolites, if applicable. 24 hours urine collection from dosing to 216 hours post-dose
Urine pharmacokinetics: percentage of dose excreted (Fe) | pre-dose and then 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  for elafibranor and metabolites, if applicable. 24 hours urine collection from dosing to 216 hours post-dose
Urine pharmacokinetics: cumulative percent of dose excreted (Fe0-t) | pre-dose and then 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  for elafibranor and metabolites, if applicable. 24 hours urine collection from dosing to 216 hours post-dose
Urine pharmacokinetics: renal clearance (CLR) | pre-dose and then 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  for elafibranor and metabolites, if applicable. 24 hours urine collection from dosing to 216 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Pascal BIRMAN, MD, Study Director — Genfit
Locations (2):
- United States (2):
  - Division of Clinical Pharmacology, University of Miami, Miami, Florida
  - inVentiv Health Clinical Research, Miami, Florida